CLINICAL TRIAL: NCT06386679
Title: A Pilot Study: Safety and Efficacy of Allogenic Mesenchymal Stem Cell Type AFCC for Treating in Elderly Knee Osteoarthritis Patients
Brief Title: Amniotic Fluid Mesenchymal Stem Cells Developed for Chondrogenic Treatment (AFCC) Injection in Elderly Knee Osteoarthritis Patients
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Tatsanee Phermthai, PhD., Principle Invesitigator, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R016634005
Record Dates: First submitted 2024-03-29; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: Amniotic fluid mesenchymal stem cells; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Ten elderly patients from both gender diagnosed with knee osteoarthritis, will be enrolled according to specific inclusion and exclusion criteria. These patients will be injected with amniotic fluid mesenchymal stem cells developed for chondrogenic treatment. Then, they are followed by clinical assessment, laboratory investigations as well as magnetic resonance imaging (MRI) of the injected knee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AFCC injection (Experimental)
  Interventions: Biological: allogenic amniotic fluid mesenchymal stem cell

INTERVENTIONS:
Biological: allogenic amniotic fluid mesenchymal stem cell — Intra-articular AFCC injection will be given for single knee for each patient in single dose, 20 million of AFCC in each dose

SUMMARY:
Amniotic fluid mesenchymal stem cells developed for chondrogenic treatment (AFCC) are used to treat elderly patients suffering from knee osteoarthritis (OA). The injection reduces inflammation and promotes the recovery of knee function, leading to an improved quality of life.

DETAILED DESCRIPTION:
Ten patients, aged between 60 and 80 of both genders, who were diagnosed with knee osteoarthritis at Kellgren and Lawrence (KL) score 2-3 were selected based on strict inclusion and exclusion criteria. Each patient was treated with a single intra-articular injection of 20 million cells of amniotic fluid mesenchymal stem cells in AFCC type into an OA knee. After the treatment, they were monitored through clinical assessment and laboratory investigation, including blood chemistry test and Magnetic Resonance Imaging (MRI) of the treated knee.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 60 to 80 years
2. The Visual Analog Scale (VAS) score of the subject's knee joint was greater than 4
3. Knee pain needs at least 15 days of experience.
4. The Kellgren Lawrence grade of the subject's knee joint was II/III as per the axial position X-ray.
5. Subjects who understand and voluntarily sign the consent.

Exclusion Criteria:

1. The subject has secondary osteoarthritis (such as other joint arthritis, major trauma on the study joint in the previous 3 months, axial deviation angle beyond 15 degrees of the bones of the knee joint)
2. The subject has other known rheumatic or inflammatory diseases (such as rheumatoid arthritis and inflammatory arthritis).
3. The subject has other conditions that cause knee joint pain (such as cancer, joint tumor)
4. The subject who awaiting knee surgery
5. The subject has an underlying disease that affects treatment during 1 year (such as cancer, liver disease, severe kidney disease, SLE)
6. The subject has a history of vertebral fracture or leg bone fracture
7. The subject has a nervous system disorder that affects balance (such as stroke or Parkinson's disease)
8. The subject has an acute or chronic infectious disease
9. The subject who had evidence of knee surgery
10. The subject who has received intra-articular steroids or other substances within the last 6 months.
11. The subject who has received symptomatic slow-acting drugs for osteoarthritis (SYSADOA) within the last 4 months
12. The subject has a deformity of the knee joint.
13. The subject has any other pathological conditions
14. The subject has a communication problem
15. The subject has claustrophobia
16. The subject who had surgery to insert a cardiac pacemaker
17. The subject who had surgery to insert an aneurysm clip
18. The subject who had surgery to insert a cochlear implant
19. The subject has any internal metallic objects (such as metal plates, surgical clips, bullets)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of abnormal physical examination | Month -3, Day 0, Month 3, 6 and 12
  The following examinations will be conducted: general appearance, respiratory, abdomen, nervous system, muscoskeletal system and etc. In case of abnormal conditions, they shall be recorded as an adverse event.
Incidence of abnormal vital sign | Month -3, Day 0, Month 3, 6 and 12
  The following assessment will be conducted: heart rate, blood pressure and temperature. In case of abnormal results, they shall be record as an adverse event.
Incidence of abnormal laboratory test results | Day 0, Month 3, 6 and 12
  The following lab tests will be conducted: serum chemistry, haematology, liver function test. In case of abnormal results, they shall be recorded as an adverse event.
Incidence of abnormal ECG parameters | Day 0, Month 3, 6 and 12
  The following assessments will be conducted: 12 lead ECG recordings with long Lead II, and two-dimensional echocardiography (2D ECHO; if needed). In case of abnormal conditions, they shall be recorded as an adverse event
The type of Adverse event (AE), numbers of AE and proportion of patients with AE. | Day 0 to 7, 14, 30, Month 2 to 12
  AE will be monitored and recorded by the investigator throughout the study.

SECONDARY OUTCOMES:
Pain score | Screening (Month -3), Day 0, Month 3, 6, and 12
  Change in pain in the affected knee joint in response to treatments using the Visual Analog Score (VAS)
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Screening (Month -3), Day 0, Month 3, 6, and 12
  Assessment changes of knee complaints by using the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
Degree of cartilage change | Screening (Month -3), Day 0, Month 3, and Month 12
  Assessment change of joint narrowing space width using Radiography (X-ray) and Magnetic Resonance Imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Tatsanee Phermthai, PhD., Study Director — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand